CLINICAL TRIAL: NCT05323968
Title: Diagnostic Accuracy of Ultrasonography and Computed Tomography in the Diagnosis of Mild-moderate Acute Diverticulitis: Prospective Cohort Study
Brief Title: Diagnostic Accuracy of Ultrasonography and Computed Tomography in the Diagnosis of Mild-moderate Acute Diverticulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Granollers (Other)
Responsible Party: Principal Investigator, Josep Maria Badia, Prof, Hospital de Granollers
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HGG2017_3
Record Dates: First submitted 2022-04-05; First posted 2022-04-12 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Acute Diverticulitis
Keywords: Ultrasonography; Computed tomography; Accuracy; Sensitivity and specifity
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Cohort study with comparison of two different diagnostic tools
Masking Description: The two imaging examinations will be done by different radiologists blinded for the previous results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acute diverticulitis (Other): Patients with clinical suspicion of acute diverticulitis
  Interventions: Diagnostic Test: Abdominal Ultrasonography; Diagnostic Test: Abdominal Computerized Tomography

INTERVENTIONS:
Diagnostic Test: Abdominal Ultrasonography — The result of the Abdominal Ultrasonography will be compared with that of the Abdominal Computerized Tomography
Diagnostic Test: Abdominal Computerized Tomography — The result of the Abdominal Computerized Tomography will be compared with that of the Abdominal Ultrasonography

SUMMARY:
Acute diverticulitis (AD) is the most common complication of diverticulosis and is divided into mild-moderate and complicated. Imaging methods are needed for its diagnosis, prognostic classification and therapeutic management. Currently the "gold-standard" imaging technique is computed tomography (CT) and most guidelines recommend it to classify and identify those patients with risk of treatment failure.

In this styudy, a prospective comparison of CT and abdominal ultrasound is proposed, with the aim of evaluating the diagnostic accuracy of ultrasound. An accurate ultrasound classification of AD would allow the differentiation of mild-moderate and complicated DA, avoiding routine CT and, therefore, patient's x-ray exposure.

DETAILED DESCRIPTION:
Study design, setting and patients. Pragmatic prospective cohort study comparing the diagnostic accuracy of US and CT scan.

During a 17-month period patients referred to the imaging department with a clinical suspicion of acute LCD will be evaluated with US and CT.

Following the hospital care protocol, patients with suspected uncomplicated LCD will first undergo an abdominal US examination. Immediately after US examination, patients will be evaluated with CT.

In emergency cases in which complicated diverticulitis is suspected, the study will start with a CT, followed by ultrasound.

The interval between both exploration test will be in all cases less than 1 hour and will be performed before the administration of any anti-inflammatory or antibiotic treatment.

US and CT exams will be performed by three different radiologists with blinded results between them. All participating radiologists have more than five years of experience in abdominal radiology.

US examinations will be performed with a scanner Aplio 500 (Canon, Tokyo, Japan) employing convex and lineal transducer. CT studies will be performed on 6-MDCT scanner (SOMATOM Emotion Siemens, Germany) following the administration of 120ml of intravenous contrast.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of acute diverticulitis

Exclusion Criteria:

* Hemodynamic instability that prevents a diagnostic delay
* Pregnant patients
* Previous history of allergy to iodinated contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Number of partcipants dignosed of having acute diverticulitis by Ultrasonography | First day of admission
  Identical imaging criteria for the diagnosis of acute diverticulitis will be used used , regardless of the image technique (US or CT).
  Following the Neff modified classification, the minimum findings to take in to account will bethe presence of diverticula and mural thickening, alone or associated with inflammation of the pericolic fat (Stage 0). Mural thickening will be considered when colonic wall has 4mm or more. Other findings will be: localized pneumoperitoneum depicted by air bubbles (Stage Ia), and abscess < 4cm (Stage Ib). Stage Ia and Ib will be considered as locally complicated diverticulitis. Findings considered as belonging to complicated diverticulitis will be: pelvic abscess > 4cm (Stage II), an intra-abdominal abscess outside the pelvis (Stage III), or difuse pneumoperitoneum and intra-abdominal free liquid (Stage IV).
Number of partcipants dignosed of having acute diverticulitis by Computerized Tomography | First day of admission
  Identical imaging criteria for the diagnosis of acute diverticulitis will be used used , regardless of the image technique (US or CT).

SECONDARY OUTCOMES:
Need of surgical operation | During admission
  Number of patients who undergo a surgical operation due to acute diverticulitis
Need of a secong evaluation by diagnostic imaging (ultrasonography or computerized tomography) | During admission
  Number of patients not improving their clinical status during treatment and need a second image evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- Fundació Privada Hospital Asil de Granollers, Granollers, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No